CLINICAL TRIAL: NCT01860742
Title: Carcinoid Tumors After Failure of Somatostatin Analogs: a Randomized Phase III of Octreotide Lutate Peptid Receptor Radionuclide Therapy (PRRT) Versus Interferon α-2b
Brief Title: Randomized Phase III of PRRT Versus Interferon
Acronym: CASTOR
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IJBMNCASTOR; 2012-005545-20 (EudraCT Number)
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Gastro-intestinal Neuroendocrine Tumors
Keywords: Peptide Receptor Radionuclide Therapy (PRRT); Neuroendocrine Tumors; Interferon alpha
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Introns; lutetium Lu 177 dotatate; 177Lu-octreotate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interferon alpha-2b (Active Comparator): Interferon α-2b in a dose of 5000000 Units administered subcutaneously every second day until progression or unacceptable adverse event from a clinical or a patient point of view.
  Interventions: Drug: Interferon alpha-2b
- 177Lu-DOTATATE (Active Comparator): intravenous injection of 177Lu-octreotate with simultaneous infusion of an aminoacid solution
  Interventions: Drug: 177Lu-DOTATATE

INTERVENTIONS:
Drug: Interferon alpha-2b — Interferon α-2b in a dose of 5000000 Units administered subcutaneously every second day
  Other Names: Intron A
  Arms: Interferon alpha-2b
Drug: 177Lu-DOTATATE — 177Lu-octreotate infusions in fixed activities of 7,4 GigaBecqurel each, given 8-11 weeks apart, injected intravenously with simultaneous infusion of an amino acid solution
  Other Names: 177Lu-octreotate; Lutate
  Arms: 177Lu-DOTATATE

SUMMARY:
The purpose of this study is to assess the benefit of 177Lu-DOTATATE versus interferon α-2b in patients with progressive, unresectable, non-pancreatic gastrointestinal neuroendocrine tumors resistant to therapy with somatostatin analogues, in terms of disease control.

DETAILED DESCRIPTION:
This is a phase III study of Peptid Receptor Radionuclide Therapy (PRRT) with 177Lu-DOTATATE versus Interferon α-2b.

Objectives of the study:

1. To assess the benefit of 177Lu-DOTATATE versus interferon α-2b in patients with progressive, unresectable,non-pancreatic gastrointestinal neuroendocrine tumors, resistant to therapy with somatostatin analogues, in terms of disease control.
2. To assess efficacy and safety parameters of both treatment arms and the predictive value of tumor 68Ga-DOTATATE PET/CT and 18FDG PET/CT uptake at baseline, at mid (+/- 16th week) and end (+/- 32th week) of treatment in both arms.

In the interferon arm: 5000000 Units of interferon will be administered subcutaneously preferentially in the evening three times a week (every other day) until disease progression.

In the 177Lu-octreotate arm: Treatment will consist of 177Lu-DOTATATE intravenous injections fractionated in fixed activities of 7,4 GigaBecquerel (200mCi) (+/- 5%), given every 8 (+/- 1) weeks with simultaneous nephroprotective infusion of an amino acid solution. (Before amino acid nephroprotection solution, ondansetron, methylprednisolone and metoclopramid, are given in infusions in order to prevent nausea or vomiting). Approximately 30 min after the beginning of the aminoacid solution, 177Lu-octreotate is injected via a second side-line over 15-30 minutes. The amino acid infusion is continued at the same rate until end (total infusion time: 4-6 hours).

In total, 4 injections of 177Lu-DOTATATE are planned. However, in respect of the absorded dose limits of critical organs(kidneys and bone marrow), the 4th 177Lu-DOTATATE injection will be tailored with a minimal administered activity of 4,6 GigaBecquerel.

Treatment efficacy will be assessed on a patient-basis using RECIST 1.1 and by Progression Free Survival. The value of tumor 68Ga-DOTATATE PET/CT and 18FDG PET/CT uptake as predicting imaging biomarkers will also be assessed in both arms.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 yrs).
2. Histology-proven non-pancreatic gastrointestinal NETs.
3. Disease progression under SSAs (SSAs-resistant disease). Disease progression must be documented with at least one of the following:

   * Radiological disease progression (according to RECIST 1.1) on an MRI or CT over the last 12 months.
   * Disease progression on a somatostatin receptor-imaging (PET/CT or SPECT/CT) over the last 12 months (apparition of new lesion(s) or increase in the transaxial plane diameter of more than 30% on the same imaging modality).
4. There should be at least one target lesion. A target lesion should fulfill all the following criteria:

   * Uptake higher than the physiological liver uptake on the baseline 68Ga-DOTATATE PET/CT
   * Longest transaxial plane diameter ≥ 20mm measured on the CT or MRI;
   * Not previously irradiated.
5. Long-acting SSAs must be discontinued at least 4 weeks before the study treatment start date and, if needed, switched to short-acting analogues which must be stopped 48h before the treatment date.
6. Adequate renal function with GFR ≥ 50 mL/min/1.73m2 (evaluated by 51Cr-EDTA test).
7. Adequate bone marrow function with:

   * Hemoglobin ≥ 9 g/dL;
   * Neutrophil ≥ 1.5·109/L;
   * Platelet count ≥ 100·109/L.
8. Adequate liver function with:

   * Total Bilirubin ≤ 2xULN;
   * Transaminases (AST and ALT) ≤ 5xULN;
   * Serum albumin > 3.0 g/dL with normal prothrombin time (>70%) unless for patients under coumarin anticoagulation therapy.
9. ECOG Performance Status ≤ 1.
10. Women of childbearing potential and men with partners of childbearing potential must agree to use a highly effective form of contraception for the duration of study participation and up to six months after the end of the treatment. A pregnancy test (serum) must be performed within 2 weeks prior to inclusion for every female patient of childbearing potential and it must be negative.
11. Patient's written informed consent obtained prior to any study specific procedure.
12. All necessary baseline procedures should be performed within 2 weeks prior to randomization date.

Exclusion Criteria:

1. Resectable tumor with curative intent.
2. Any major surgery within the last 6 weeks prior to inclusion in the study.
3. Radiotherapy, chemotherapy, embolization, mammalian target of rapamycin (mTOR)-inhibitors, receptor tyrosine-kinase inhibitors or other investigational therapy within 12 weeks prior to inclusion in the study.
4. Previous PRRT or MIBG treatment.
5. Treatment with interferon 12 months prior to inclusion in the study.
6. Presence of non-benign 18FDG-positive lesions (higher than 2 x normal liver (or thoracic aorta uptake -SUVmax- in case of liver involvement)) without significant 68Ga-DOTATATE uptake.
7. Uncontrolled congestive heart failure (NYHA stade ≥ 2).
8. Diffuse bone marrow infiltration on the baseline 68Ga-DOTATATE PET/CT confirmed by MRI.
9. Prior external beam radiotherapy on kidneys or on more than 25% of bone marrow.
10. Patients with known uncontrolled brain metastases.
11. History of other active malignant disease or clinical remission less than 5 years (except in case of non melanoma skin cancer or in situ cervical carcinoma).
12. Known autoimmune hepatitis.
13. Patients after organ transplantation under immunosuppressive therapy.
14. Patients with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the investigator's opinion, may interfere with completion of the study.
15. Hypersensitivity to interferon α-2b or to any component of the product.
16. Pregnant or lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 3 years [Anticipated]
  PFS is defined by the time between treatment initiation and the first of the following events:
  * Disease progression according to RECIST 1.1;
  * Death of the patient from any cause;
  * Appearance of confirmed new lesion(s) on 68Ga-DOTATATE PET/CT or 18FDG PET/CT.

SECONDARY OUTCOMES:
Treatment response according to RECIST 1.1 (Response Evaluation Criteria In Solid Tumors) | 3 years [Anticipated]
Adverse events according to Common Terminology Criteria for Adverse Events version 4.03 (CTC 4.03-WHO criteria) | 3 years [Anticipated]
Tumor 18FDG PET/CT and 68Ga-octreotate PET/CT uptake at baseline, at mid and end of treatment | 3 years [Anticipated]

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Flamen, M.D., Ph.D., Principal Investigator — Jules Bordet Institute; Christophe Deroose, M.D., Ph.D., Principal Investigator — UZ Leuven
Locations (2):
- Belgium (2):
  - Jules Bordet Institute, Brussels
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No